CLINICAL TRIAL: NCT04271137
Title: Evaluation of Orbital Reconstruction Using Patient Specific 3-D Printed Onlay Versus Pre-Bent Titanium Mesh
Brief Title: Correction of Enophthalmos and Orbital Volume Using Pre-bent Mesh Versus 3d Printed Onlay in Orbital Fracture Cases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Salah, Principal investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMFS 3 3 10
Record Dates: First submitted 2020-02-10; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Orbital Fractures; Enophthalmos; Periorbital Fracture
Keywords: 3d printed onlay; PEEK; orbital mesh; computer-guided surgery
MeSH Terms: conditions — Orbital Fractures; Enophthalmos

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Orbital fractues (Other): Orbital fractures
  Interventions: Combination Product: 3D printed PEEK onlay; Combination Product: Pre-bent orbital mesh

INTERVENTIONS:
Combination Product: 3D printed PEEK onlay — 3d computer-designed Orbital onlay
Combination Product: Pre-bent orbital mesh — Pre-bent orbital mesh on 3d printed template

SUMMARY:
this study evaluates the post-surgical correction of enophthalmos and orbital volume using 3D printed only versus pre-bent titanium mesh in blow-out fracture cases

DETAILED DESCRIPTION:
Many materials had been used in reconstruction of blow out fractures, the aim of this study is to evaluate the enophthalmos correction and orbital volume restoration using 3D printed onlay versus pre-bent titanium mesh

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≤17 years old).
* Blow-out Orbital Fracture.
* Unilateral Orbital Trauma.
* Enophthalmos (≤ 2 mm).
* Patients with contralateral healthy, non-surgically operated orbit.

Exclusion Criteria:

* Young Patients (> 17 years old).
* Patients with Systemic diseases.
* Bilateral Orbital Trauma.
* Enophthalmos (>2 mm).
* Patients whom cannot tolerate follow up intervals.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Enophthalmos | 1 week post-operative
  CT based exphthalmometery - corneal projection from lateral orbital rim measured in millimeters
Enophthalmos | 1 year post-operative
  CT based - corneal projection from lateral orbital rim measured in millimeters

SECONDARY OUTCOMES:
Orbital volume | one week post-operative
  Change in orbital volume ratio on CT in centimeter cubic
Implant position accuracy | One week post-operative
  Superimposition of pre- and post-operative 3d bony structures on CT in 2d views of the x-ray

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mohamed, PhD, Study Director — Cairo University
Locations (1):
- Faculty of Dentistry - Cairo University, Cairo, Egypt